CLINICAL TRIAL: NCT02764216
Title: Elective Mucosal Irradiation in Head-and Neck Cancer of Unknown Primary, A Single Arm Phase II Trial
Brief Title: Elective Mucosal Irradiation in Head-and-Neck Cancer of Unknown Primary
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guopei Zhu, M.D., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1501160-4
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Head-and-neck Cancer; Carcinoma of Unknown Primary
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms, Unknown Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EMI group (Experimental): Elective mucosal irradiation
  Interventions: Radiation: Elective mucosal irradiaton

INTERVENTIONS:
Radiation: Elective mucosal irradiaton — Patients will elective mucosal irradiaton based on nodal station, EBV/HPV status, RPN status etc. IMRT will be adopted.

SUMMARY:
The optimal treatment of HNCUP remains controversial and lacks evidence from prospective randomized trials. The management of these patients relies primarily on surgery and radiotherapy. The role of radiotherapy in sterilizing putative mucosal sites remains controversial. The main debate concerns the extent of the radiation field. Although pan-mucosal irradiation from the nasopharynx to the hypopharynx and bilateral neck nodes reduces the risk of emergence of a mucosal primary or a nodal relapse, it has been associated with significant toxicity and long-term morbidity (mostly xerostomia and dysphagia). Most single institution retrospective studies have not shown any advantage for more extensive irradiation.Therefore, elective mucosal irradiation may might be appropriate only for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Carcinomas metastatic to cervical lymph node with unknown primary
2. Squamous cell carcinoma, poorly differentiated carcinoma, or undifferentiated carcinoma
3. All patients must be suitable to attend regular follow-up and undergo toxicity assessment.
4. Stage T0, N1-3, M0 disease
5. Karnofsky score over 60
6. No significant cardiac, chest, gastrointestinal or renal morbidities

Exclusion Criteria:

1. Previous radiotherapy to the head and neck region
2. Previous malignancy except non-melanoma skin cancer
3. Previous or concurrent illness which in the investigators opinion would interfere with either completion of therapy or follow-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2010-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Mucosal recurrence free survival | 3 years
  from date of enrollment to date of first documented primary site emergence or death, assessed up to 3 years.

SECONDARY OUTCOMES:
Disease-free survival | 3 years
  from date of enrollment until date of first documented disease progression or death from any cause, assessed up to 3 years.
Neck control rate | 3 years
  from date of enrollment until date of first documented neck relapse, assessed up to 3 years.
overall survival rate | 3 years
  from date of enrollment until date of first death from any cause, assessed up to 3 years.
Acute toxicities(gastrointestinal toxicities,hematologic toxicities, dysphagia,oral mucositis) | 2 months
  Acute toxicities(gastrointestinal toxicities,hematologic toxicities, dysphagia,oral mucositis) during the course of radiotherapy

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai ninth people's hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dou S, Li R, Zhang L, Wang Z, Xie L, Zhang C, Zhu G. Long-term results of elective mucosal irradiation for head and neck cancer of unknown primary in Chinese population: The EMICUP study. Cancer Med. 2020 Mar;9(5):1712-1720. doi: 10.1002/cam4.2856. Epub 2020 Jan 17. PMID 31953927